CLINICAL TRIAL: NCT04800263
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of Single Subcutaneous Administered SHR-1905 in Healthy Subjects
Brief Title: A Trial of SHR-1905 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-1905-I-101-AUS
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SHR-1905 Dose Level 1 (Experimental): SHR-1905 Dose level 1
  Interventions: Drug: SHR-1905; Drug: Placebo
- SHR-1905 Dose Level 2 (Experimental): SHR-1905 Dose level 2
  Interventions: Drug: SHR-1905; Drug: Placebo
- SHR-1905 Dose Level 3 (Experimental): SHR-1905 Dose level 3
  Interventions: Drug: SHR-1905; Drug: Placebo
- SHR-1905 Dose Level 4 (Experimental): SHR-1905 Dose level 4
  Interventions: Drug: SHR-1905; Drug: Placebo
- SHR-1905 Dose Level 5 (Experimental): SHR-1905 Dose level 5
  Interventions: Drug: SHR-1905; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1905 — SHR-1905 will be injected subcutaneously
Drug: Placebo — Placebo will be injected subcutaneously

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single dose escalation phase 1 study. The objective of this study is to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of subcutaneous administered SHR-1905 in healthy subjects.

DETAILED DESCRIPTION:
The study will consist of one dose esclation part with a total of 5 dose levels. The Subjects will be randomized to receive SHR-1905 as reflected by the guiding principle for the dose esclation/expansion phase. Each dose group includes a screening period, a baseline period, an observational period, and a safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, volunteers to participate in the trial.
2. Male or female aged between 18 years and 55 years (inclusive) at the date of signed consent form.
3. Total body weight ≥45 kg at screening, and body mass index (BMI) between 18 and 28 kg/m2 (inclusive).
4. For healthy subjects, no clinically significant abnormalities.
5. Men and women of childbearing potential (WOCBP) must agree to take effective contraceptive methods

Exclusion Criteria:

1. Known medical history of severe disease in cardiovascular, liver, kidney, digestive tract, mental nerve, hematology, metabolic disorders, etc.
2. Severe injuries or major surgeries within 6 months before screening.
3. Subjects with infecious disease.
4. Hyper/Hypotension at screening and at check in.
5. Clinically significant abnormalities in 12-Lead ECG
6. More than 5 cigarettes daily (or products with equivalent amount of nicotine) for 3 months prior to screening
7. Positive urine drug screen .
8. Subject who cannot perform venous blood sampling.
9. Known history or suspected of being allergic to the study drugs and their excipients.
10. Use of any medicine within 4-weeks or within 5 half-lives
11. History of alcohol abuse within 3 months prior to the IP administration .
12. Participation in clinical trials of other investigational drugs or medical devices within 3 months prior to screening
13. in the investigator's judgment, may increase the risk to the subject

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 16 weeks)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (approximately 16 weeks)
  Area under the concentration-time curve from time 0 to last time point after SHR-1905 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 16 weeks)
  Area under the concentration-time curve from time 0 to infinity after SHR-1905 administration
Pharmacokinetics-Tmax | Start of Treatment to end of study (approximately 16 weeks)
  Time to Cmax of SHR-1905
Pharmacokinetics-Cmax | Start of Treatment to end of study (approximately 16 weeks)
  Maximum observed concentration of SHR-1905
Pharmacokinetics-CL/F | Start of Treatment to end of study (approximately 16 weeks)
  Apparent clearance of SHR-1905
Pharmacokinetics-Vz/F | Start of Treatment to end of study (approximately 16 weeks)
  Apparent volume of distribution during terminal phase of SHR-1905
Pharmacokinetics-t1/2 | Start of Treatment to end of study (approximately 16 weeks)
  Terminal elimination half-life of SHR-1905
Anti-Drug antibody | Start of Treatment to end of study (approximately 16 weeks)
  The percentage of subjects with positive ADA titers over time for SHR-1905

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fei Y, Li N, Qian W, Fan Y, Shen Y, Wang Q, McLendon K, Shen K. A phase 1, randomized, double-blind, placebo-controlled, dose escalation study to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of SHR-1905, a long-acting anti-thymic stromal lymphopoietin antibody, in healthy subjects. Front Pharmacol. 2024 Jul 15;15:1400696. doi: 10.3389/fphar.2024.1400696. eCollection 2024. PMID 39076593